CLINICAL TRIAL: NCT03486002
Title: EFFECTS OF TELEFLEX CATHETER (CLEANSWEEP) ON VENTILATOR MECHANICS
Brief Title: EFFEXTS OF THE CLEANSWEEP SUCTION CATHETER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Access to the devices was halted by the sponsor
Sponsor: Duke University (Other)
Collaborators: Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00087066
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2019-09

CONDITIONS: Endotracheal Tube Clearance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cleansweep closed suction system (Other)
  Interventions: Device: Cleansweep
- Halyard closed suction system (Other)
  Interventions: Device: Halyard

INTERVENTIONS:
Device: Cleansweep — The Cleansweep closed suction system
  Arms: Cleansweep closed suction system
Device: Halyard — Halyard Closed Suction System
  Arms: Halyard closed suction system

SUMMARY:
This study is designed to compare the effectiveness of a closed suction system with an inflatable balloon on the catheter (Cleansweep system) to that of a standard closed suction system in terms of reducing the interior resistance of endotracheal tubes. Subjects who require frequent suctioning ( > every 2.5 hours) and who have stable cardiovascular systems will be randomized to receive suctioning either through the Cleansweep system or standard system initially followed by the corresponding system. The subjects will be suctioned every two hours for eight hours ( the first 2 suction procedures with one system followed by 2 with the other system). After each suction procedure measurements of resistance will be made using peak and plateau pressures.

Analysis: For each patient, data for both procedures on each catheter system will be pooled and mean differences between the standard system and the Cleansweep system will be calculated. For all 20 patients the mean (+/- SD) of these differences will be calculated and significance will be sought using appropriate statistical tests. The study will be unblinded and randomization determines merely which system will used initially for the first 2 procedures.

ELIGIBILITY:
Inclusion Criteria:

* Intubated, mechanically ventilated patients who require suctioning more often than every 2.5 hours

Exclusion Criteria:

* Unstable cardiovascular system (significant arrythmias, blood pressure support requiring > 2 pressors
* refractory hypoxemia (P/F ratio < 80)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Change in endotracheal tube resistance during mechanical ventilation after 4 suction procedures | 8 hours
  Measurements of resistance will be made following each suction procedure (2 with the Cleansweep system and 2 with the standard system)

CONTACTS AND LOCATIONS:
Overall Officials: Neil MacIntyre, Principal Investigator — Duke University
Locations (1):
- Duke Health System, Durham, North Carolina, United States